CLINICAL TRIAL: NCT04089332
Title: Insulin Resistance, Cognitive Health, and Perfusion of the Adolescent Brain
Brief Title: Insulin Resistance in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2019-0361; 1R21HD097510-01A1 (NIH); A176000 (Other: UW Madison); EDUC/KINESIOLOGY/KINESIOLOG (Other: UW Madison); 19PRE34450141 (Other Grant/Funding Number: American Heart Association); Protocol Version 9/24/2021 (Other: UW Madison)
Record Dates: First submitted 2019-09-03; First posted 2019-09-13 (Actual); Results first posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Insulin Resistance
MeSH Terms: conditions — Insulin Resistance | interventions — Glucose Tolerance Test; Vascular Access Devices; Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Enrolled, eligible (Experimental): Single arm for eligible subjects
  Interventions: Other: Oral Glucose Tolerance Test (OGTT); Device: 3 Tesla MRI; Device: Intravenous Catheter; Other: Cognitive Tests

INTERVENTIONS:
Other: Oral Glucose Tolerance Test (OGTT) — Eligible subjects will undergo MRI scanning before and after oral glucose tolerance test.
  Other Names: OGTT
Device: 3 Tesla MRI — A 3 Tesla MRI will be used to assess brain structure, quantify cerebral blood flow and capture cerebral vessel structure at designated time points throughout the study visits.
  Other Names: MRI
Device: Intravenous Catheter — A blood sampling IV catheter will be used to draw blood samples at specific time points throughout each study visit to measure concentrations of glucose and insulin.
  Other Names: Cath
Other: Cognitive Tests — A battery of cognitive tests will be completed by the subject.

SUMMARY:
The growing population of adolescents with insulin resistance (IR) is predicted to create a large public health burden in the next few decades. This study examines the function of brain blood vessels and cognitive function, to test if increasing severity of IR in adolescents is related to reduced cognitive function and reduced brain blood vessel function. Findings from this study may help create treatments to delay or prevent some of the negative effects of IR on cognitive and vascular health.

DETAILED DESCRIPTION:
One in five American adolescents is obese. Up to half of those are already exhibiting insulin resistance (IR), a hallmark of metabolic syndrome and diabetes linked to serious life-altering health disorders, including cardiovascular and cerebrovascular disease. In adults, IR negatively affects brain structure and function and is reflected in lower regional brain volumes, perfusion, increased white matter hyperintensities and abnormal neuropsychological status, especially affecting memory and attention-all changes associated with accelerated cognitive and brain aging and increased risk of dementia. In an analogous fashion, a limited set of literature suggests adolescents with IR exhibit similar brain changes during maturation. The investigators hypothesize that the brains of obese adolescents are more susceptible to insults of IR during rapid brain development, positioning them on an abnormal cognitive trajectory, and predisposing them to issues related to learning, behavioral stress responses, and depression.

While the metabolic consequences of IR are well described in adolescence, the impact of IR on their neurocognitive status (intelligence, memory, attention, executive function, processing speed) and cerebrovascular function and their interactions remains largely unexplored. This is important since in addition to its classic role as a metabolic hormone, insulin acts as a vasodilator and supports neurotrophic signaling in healthy humans. Therefore, dysfunctional insulin signaling may hold tremendous influence over brain health in adolescents during this vital period of brain development. New insight is required to understand where, when, and how IR negatively transforms brain health, including whether a dose-response exists between IR severity and anomalies in brain and cognition.

The long-term goal of this research program is to determine the influence of IR on brain development in adolescents through the relationships between neurocognition and cerebral blood supply. The primary goal of the current project is to quantify fundamental neurocognitive and cerebrovascular function in relation to the severity of IR. The central hypothesis is that as IR worsens: a) subtle but meaningful neurocognitive declines emerge; b) regional brain perfusion is reduced primarily in areas linked to learning and memory despite preserved resting global cerebral blood flow (CBF); c) acute insulin surges exacerbate regional hypoperfusion, and d) cognitive scores will be lower, mediated in part by insulin-stimulated hypoperfusion.

Participants will be recruited primarily from pediatric and pediatric endocrinology clinics via our collaborator, Dr. Aaron Carrel, and his staff in UWHC Pediatric Endocrinology. Additionally, participants will be recruited from the greater Madison, WI community.

ELIGIBILITY:
Inclusion Criteria:

* Age 12-18 years inclusive
* Typically developing and cognitively intact

Exclusion Criteria:

* Diabetes (≥126 mg dL-1 fasting glucose)
* Insulin treatment or sensitizing drugs
* Diagnosis of kidney, pulmonary, or heart disease
* Current smoking (defined as use of nicotine >5 times in the past month)
* Pregnancy
* Neurological or developmental disorders (e.g., intellectual disability, autism)
* Significant head injury or medical conditions (e.g., concussion, encephalopathy, seizure disorder)
* Inability to undergo the MRI procedure
* Weight less than 94.5 lbs (42.9 kg) to adhere to safety guidelines regarding blood sampling and OGTT administration
* Tanner Stage <3
* Any other circumstance deemed by the PI not addressed above

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2019-10-04 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Schrage, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin-Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from October 2019 to April 2022. Participants were 12-18 years old during Covid-19 pandemic, and thus had very delayed access to vaccines, limiting enrollment. Pandemic related safety issues effected study conduct. Not all enrolled participants completed all (up to 5, 3 for the primary aims) study visits as a result. Because the data collected in each visit was not dependent on the other visit in a temporal manner, the study visits could occur in any order.
Pre-assignment Details: 34 participants were consented, but due to the Covid-19 pandemic, only 23 participants started the study (completed at least 1 study visit).
Groups:
- Enrolled, Eligible: Oral Glucose Tolerance Test: Eligible subjects will undergo MRI scanning before and after oral glucose tolerance test.
  3 Tesla MRI: A 3 Tesla MRI will be used to assess brain structure, quantify cerebral blood flow and capture cerebral vessel structure at designated time points throughout the study visits.
  Intravenous Catheter: A blood sampling IV catheter will be used to draw blood samples at specific time points throughout each study visit to measure concentrations of glucose and insulin.
  Cognitive Tests: A battery of cognitive tests will be completed by the subject.
Period: Overall Study
Arm/Group | Enrolled, Eligible
Started | 23
Completed Cognitive Tests | 13
Completed OGTT | 17
Completed MRI Structural Visit | 16
Completed With Data to Analyze | 15
Participants With Data for Change in CBF | 11
Completed | 15
Not Completed | 8
Not completed — COVID-19 Pandemic safety issues | 6
Not completed — Moved in the MRI, no analysis possible | 1
Not completed — Completed only OGTT, no analysis possible | 1

BASELINE CHARACTERISTICS:
Population: Demographics provided for the 15 participants for whom enough data was collected to analyze the relationship between HOMA-IR, Cognitive Abilities, and Cerebral Blood Flow.
Arm/Group | Enrolled, Eligible
Number analyzed (Participants) | 15
Age, Continuous [Mean (Full Range); unit: years] | 14.53 [12 to 18]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Linear Relationship Between HOMA-IR and Cognitive Function (R-squared)
Description: HOMA-IR was measured from each participant at baseline (up to 1 hour visit) and a battery of cognitive instruments (listed here) were measured at a different study visit (2-3 hours of time). A relationship between individual HOMA-IR and Cognitive Function was hypothesized and a measured via Linear Regression (R-squared).
Time Frame: data collected at baseline visit (HOMA-IR) and one other study visit (Cognitive Function Tests) (up to 4 hours total time of data collection over two visits - data collection not temporally dependent)
Population: This includes all the participants that completed the cognitive visit of the study. Because data collected in each visit was not dependent on other visits in a temporal manner, study visits occurred in any order.
Measure: Number; unit: R-squared
Arm/Group | Enrolled, Eligible
Number analyzed (Participants) | 13
R-squared
  WASI II (Verbal IQ) Measure of intellectual ability, sub-tests Vocabulary and Similarities | 0.205
  WASI II (Performance IQ) Measure of intellectual ability, sub-tests Block Design, Matrix Reasoning | 0.299
  NIH Toolbox (List Learning) A cognitive measure of working memory | 0.738
  NIH Toolbox (Oral Symbol Digit Test) A cognitive measure of processing speed (numbers/symbols) | 0.0264
  NIH Toolbox (Flanker Inhibitory Control and Attention) Executive function measure | 0.186
  NIH Toolbox (Pattern Comparison) A cognitive measure of processing speed (stimuli) | 0.04
  NIH Toolbox (Picture Sequence) A cognitive measure of episodic memory | 0.47
  WRAML (Picture Memory) A general memory measure of picture recognition | 0.0572
  D-KEFS (Color Word Interference) A measure of cognitive flexibility through inhibition | 0.000224
  D-KEFS (Trail Making Test) A measure of mental flexibility (motor speed) | 0.392
  Peds QL (Child 8-12 / Teen 13-18) A measure of health-related quality of life (HRQOL) in children | 0.481
Statistical Analysis 1: Comparison: Enrolled, Eligible; WASI II (Verbal IQ) vs HOMA-IR; Test type: Other; p = 0.162, Regression, Linear; Slope = -0.4465; Adjusted R-squared = 0.117
Statistical Analysis 2: Comparison: Enrolled, Eligible; WASI II (Performance IQ) vs HOMA-IR; Test type: Other; p = 0.082, Regression, Linear; Slope = 0.6704; Adjusted R-squared = 0.221
Statistical Analysis 3: Comparison: Enrolled, Eligible; NIH Toolbox (Flanker Inhibitory Control and Attention) vs HOMA-IR; Test type: Other; p = 0.286, Regression, Linear; Slope = -0.8486; Adjusted R-squared = 0.0503
Statistical Analysis 4: Comparison: Enrolled, Eligible; NIH Toolbox (Pattern Comparison) vs HOMA-IR; Test type: Other; p = 0.635, Regression, Linear; Slope = -0.0266; Adjusted R-squared = 0
Statistical Analysis 5: Comparison: Enrolled, Eligible; NIH Toolbox (Picture Sequence) vs HOMA-IR; Test type: Other; p = 0.061, Regression, Linear; Slope = -0.1588; Adjusted R-squared = 0.381
Statistical Analysis 6: Comparison: Enrolled, Eligible; WRAML (Picture Memory) vs. HOMA-IR; Test type: Other; p = 0.479, Regression, Linear; Slope = 0.099; Adjusted R-squared = 0
Statistical Analysis 7: Comparison: Enrolled, Eligible; D-KEFS (Color-Word Interference) vs. HOMA-IR; Test type: Other; p = 0.965, Regression, Linear; Slope = 0.0676; Adjusted R-squared = 0
Statistical Analysis 8: Comparison: Enrolled, Eligible; D-KEFS (Trail Making Test) vs. HOMA-IR; Test type: Other; p = 0.039, Regression, Linear; Slope = -0.0091; Adjusted R-squared = 0.324
Statistical Analysis 9: Comparison: Enrolled, Eligible; PedsQL (Child 8-12 / Teen 13-18) vs. HOMA-IR; Test type: Other; p = 0.018, Regression, Linear; Slope = -4.2085; Adjusted R-squared = 0.0423

2. Primary Outcome: Change in Cerebral Blood Flow (CBF) as Determined by MRI (mL/100g/Min)
Description: CBF will be measured via MRI before OGTT (baseline) and after OGTT at Peak insulin.
Time Frame: 1 study visit, measured at baseline and peak insulin (45-60 minutes after baseline)
Measure: Mean (Standard Deviation); unit: mL/100g/min
Groups:
- Enrolled, Eligible: Single arm for eligible subjects
  Oral Glucose Tolerance Test: Eligible subjects will undergo MRI scanning before and after oral glucose tolerance test.
  3 Tesla MRI: A 3 Tesla MRI will be used to assess brain structure, quantify cerebral blood flow and capture cerebral vessel structure at designated time points throughout the study visits.
  Intravenous Catheter: A blood sampling IV catheter will be used to draw blood samples at specific time points throughout each study visit to measure concentrations of glucose and insulin.
  Cognitive Tests: A battery of cognitive tests will be completed by the subject.
Arm/Group | Enrolled, Eligible
Number analyzed (Participants) | 11
mL/100g/min
  Perfusion of Gray Matter at Baseline | 64.25666 (11.24309)
  Perfusion of Gray Matter at Peak Insulin (Avg. 45 min) | 66.96387836 (13.93884706)
  Change in Perfusion of Gray Matter | 2.707215114 (5.642163965)
Statistical Analysis 1: Comparison: Enrolled, Eligible; Change in Gray Matter Perfusion vs. HOMA-IR; Test type: Other; p = 0.558, Regression, Linear; Slope = -1.1138; Adjusted R-square = 0
Statistical Analysis 2: Comparison: Enrolled, Eligible; Baseline Gray Matter vs. HOMA-IR; Test type: Other; p = 0.057, Regression, Linear; Slope = -5.8089; Adjusted R-squared = 0.18

3. Primary Outcome: Linear Relationship Between Cerebral Blood Flow and Cognitive Function (R-squared)
Description: Cerebral Blood Flow was measured from each participant at baseline (without OGTT MRI Visit) and a battery of cognitive instruments (those listed below) were measured at a different study visit. A relationship between individual Cerebral Blood Flow and Cognitive Function was hypothesized and a measured via Linear Regression (R-squared).
Time Frame: data collected at baseline (CBF - up to 1 hour) and Cognitive Function data collected at another study visit (up to 3 hours), data collection over 2 study visits up to 4 hours total, data collection not temporally dependent
Population: as for outcome 1
Measure: Number; unit: R-squared
Arm/Group | Enrolled, Eligible
Number analyzed (Participants) | 13
R-squared
  WASI II (Verbal IQ) Measure of intellectual ability, sub-tests Vocabulary and Similarities. | 0.132
  WASI II (Performance IQ) Measure of intellectual ability, sub-tests Block Design, Matrix Reasoning | 0.119
  NIH Toolbox (List Learning) A cognitive measure of working memory | 0.06
  NIH Toolbox (Oral Symbol Digit Test) A cognitive measure of processing speed (numbers/symbols) | 0.0593
  NIH Toolbox (Flanker Inhibitory Control and Attention) Executive function measure | 0.366
  NIH Toolbox (Pattern Comparison) A cognitive measure of processing speed (stimuli) | 0.000497
  NIH Toolbox (Picture Sequence) A cognitive measure of episodic memory | 0.0688
  WRAML (Picture Memory) A general memory measure of picture recognition | 0.185
  D-KEFS (Color-Word Interference) A measure of cognitive flexibility through inhibition | 0.234
  D-KEFS (Trail Making Test) A measure of mental flexibility (motor speed) | 0.00466
  PedsQL (Child 8-12 / Teen 13-18) A measure of health-related quality of life (HRQOL) in children | 0.0344
Statistical Analysis 1: Comparison: Enrolled, Eligible; WASI II (Verbal IQ) vs. Cerebral Blood Flow; Test type: Other; p = 0.377, Regression, Linear; Slope = -0.4465; Adjusted R-squared = 0
Statistical Analysis 2: Comparison: Enrolled, Eligible; WASI II (Performance IQ) vs. Cerebral Blood Flow; Test type: Other; p = 0.402, Regression, Linear; Slope = 0.6704; Adjusted R-squared = 0
Statistical Analysis 3: Comparison: Enrolled, Eligible; NIH Toolbox (Flanker Inhibitory Control and Attention) vs. Cerebral Blood Flow; Test type: Other; p = 0.203, Regression, Linear; Slope = -0.8486; Adjusted R-squared = 0.207
Statistical Analysis 4: Comparison: Enrolled, Eligible; NIH Toolbox (Pattern Comparison) vs. Cerebral Blood Flow; Test type: Other; p = 0.967, Regression, Linear; Slope = -0.0266; Adjusted R-squared = 0
Statistical Analysis 5: Comparison: Enrolled, Eligible; NIH Toolbox (Picture Sequence) vs. Cerebral Blood Flow; Test type: Other; p = 0.616, Regression, Linear; Slope = -0.1588; Adjusted R-squared = 0
Statistical Analysis 6: Comparison: Enrolled, Eligible; WRAML (Picture Memory) vs. Cerebral Blood Flow; Test type: Other; p = 0.287, Regression, Linear; Slope = 0.099; Adjusted R-squared = 0.0497
Statistical Analysis 7: Comparison: Enrolled, Eligible; D-KEFS (Color-Word Interference) vs. Cerebral Blood Flow; Test type: Other; p = 0.225, Regression, Linear; Slope = 0.0676; Adjusted R-squared = 0.106
Statistical Analysis 8: Comparison: Enrolled, Eligible; D-KEFS (Trail Making Test) vs. Cerebral Blood Flow; Test type: Other; p = 0.872, Regression, Linear; Slope = -0.0091; Adjusted R-squared = 0
Statistical Analysis 9: Comparison: Enrolled, Eligible; PedsQL (Child 8-12 / Teen 13-18) vs. Cerebral Blood Flow; Test type: Other; p = 0.66, Regression, Linear; Slope = -4.2085; Adjusted R-squared = 0

4. Primary Outcome: Mediation Analysis of the Indirect Effect of Cerebral Blood Flow on Insulin Resistance and Cognitive Function
Description: Mediation analysis is a statistical method used to explain the influence of an outside variable (mediator) that may modify the direct relationship between the Independent (X) and Dependent variable (Y).
  (X - Mediator - Y)
  Mediation analysis was used to explore the impact of cerebral blood flow on the relationship between HOMA-IR and cognitive function. This analysis was conducted on 11 separate cognitive function tests, looking at verbal skills, memory, executive function, and self-reported quality of life rating. In the first set of analyses, the mediator was "grey matter baseline", which is the cerebral blood flow in the resting state. The second set of analyses, the mediator was "grey matter change with OGTT", which is the cerebral blood flow changing from rest to response from Oral Glucose Tolerance Test (OGTT).
  Positive/negative effect numbers indicated that the total effect of the relationship was positive/negative.
Time Frame: through study completion (up to 2 years)
Population: Mediation analysis was conducted on a limited data set due to the low number of participants.
Measure: Number; unit: beta value
Arm/Group | Enrolled, Eligible
Number analyzed (Participants) | 13
beta value
  HOMA-IR vs WASii- Verbal (Grey Matter Baseline) | 1.6787
  HOMA-IR vs WASii-Performance (grey Matter Baseline) | -3.3431
  HOMA-IR vs WRAML (Grey Matter Baseline) | -0.8194
  HOMA-IR vs DKEFS Trail Making (Grey Matter Baseline) | -0.1702
  HOMA-IR vs DKEFS Inhibition Stroop (Grey Matter Baseline) | -0.2095
  HOMA-IR vs PEDS QL Child Report (Grey Matter Baseline) | 30.7925
  HOMA-IR vs NIH Toolbox Verbal List Learning (Grey Matter Baseline) | 0.5834
  HOMA-IR vs NIH Toolbox Oral Digit Symbol (Grey Matter Baseline) | 6.98
  HOMA-IR vs NIH Toolbox Flanker (Grey Matter Baseline) | 1.0747
  HOMA-IR vs NIH Toolbox Pattern Comparison (Grey Matter Baseline) | 2.3718
  HOMA-IR vs NIH Toolbox Picture Memory (Grey Matter Baseline) | -0.9954
  HOMA-IR vs WASii- Verbal (Grey Matter Change with OGTT) | -0.9125
  HOMA-IR vs WASii-Performance (grey Matter Change with OGTT) | -2.8222
  HOMA-IR vs WRAML (Grey Matter Change with OGTT) | -0.0008
  HOMA-IR vs DKEFS Trail Making (Grey Matter Change with OGTT) | 0.1719
  HOMA-IR vs DKEFS Inhibition Stroop (Grey Matter Change with OGTT) | -0.3754
  HOMA-IR vs PEDS QL Child Report (Grey Matter Change with OGTT) | -7.4081
  HOMA-IR vs NIH Toolbox Verbal List Learning (Grey Matter Change with OGTT) | 0.2067
  HOMA-IR vs NIH Toolbox Oral Digit Symbol (Grey Matter Change with OGTT) | -2.1898
  HOMA-IR vs NIH Toolbox Flanker (Grey Matter Change with OGTT) | -2.8883
  HOMA-IR vs NIH Toolbox Pattern Comparison (Grey Matter Change with OGTT) | 0.5842
  HOMA-IR vs NIH Toolbox Picture Memory (Grey Matter Change with OGTT) | -1.5724

ADVERSE EVENTS:
Time Frame: up to 1 year and 9 months (this was the longest any one participant was on study)
Arm/Group | Enrolled, Eligible
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 2/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled, Eligible (N=23)
Unrelated Broken Bone (General disorders) | 1 (1) — Subject dislocated left patella, not at study visit.
Unrelated Hip Injury (General disorders) | 1 (1) — Subject reported sports-related hip injury approximately 1-month prior. Physician evaluated with no intervention.

LIMITATIONS AND CAVEATS:
Study conduct was impacted by the COVID-19 pandemic. Safety issues with the target population during this time influenced whether participants completed any or all of the study visits.

Due to the small sample size, the statistic tests are likely underpowered and should be interpreted with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-24): https://cdn.clinicaltrials.gov/large-docs/32/NCT04089332/Prot_SAP_000.pdf